CLINICAL TRIAL: NCT05273216
Title: Hemodynamic Changes and Reperfusion Injury After Endovascular Stroke Treatment: Prospective Multicenter DYNASTROKE STUDY
Brief Title: Reperfusion Injury After Endovascular Stroke Treatment
Acronym: DYNASTROKE
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: Medical University Innsbruck (Other); Paracelsus Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: EK 30-254 ex 17/18
Record Dates: First submitted 2022-02-15; First posted 2022-03-10 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Ischemic Stroke
Keywords: Endovascular Stroke Treatment; Mechanical Thrombectomy; Reperfusion Injury; Intracranial Hemorrhage; Transcranial Duplex Sonography; Perfusion MRI; Cerebral Hyperperfusion
MeSH Terms: conditions — Ischemic Stroke; Reperfusion Injury; Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Study (no different study arms): Prospective, longitudinal, multicenter, observational study to investigate hemodynamic changes (by TCD and perfusion MRI) and blood biomarkers as predictors of reperfusion injury / intracranial hemorrhage after stroke thrombectomy of the anterior cerebral circulation
  Interventions: Diagnostic Test: Transcranial Duplex Sonography; Diagnostic Test: Brain MRI; Diagnostic Test: Blood biomarkers

INTERVENTIONS:
Diagnostic Test: Transcranial Duplex Sonography — Immediately after mechanical thrombectomy, patients will be investigated with bedside neurosonography (including TCD) at the stroke unit or neurointensive care unit. Apart from routine assessment of brain-supplying vessels, experienced sonographers will especially focus on intracranial blood flow velocities and determine the MCA mean blood flow velocity index (recanalized divided by contralateral artery). To assess potential dynamic blood flow changes, these investigations will be repeated at 24-48 hours after thrombectomy and at day 7 when we expect a (more) stable stroke phase. During these neurosonographic assessments, other important and potentially influential (hemodynamic) parameters such as blood pressure, heart rate and use of vasoactive medications will be documented. Assessment of intracranial blood flow will be standardized to dedicated measuring points.
Diagnostic Test: Brain MRI — The investigators will use magnetic resonance imaging (MRI) and magnetic resonance angiography (MRA) routinely performed on day 1 after thrombectomy to assess (1) the size and location of acute ischemic damage including (vasogenic) cerebral edema formation, (2) hemorrhagic transformation, (3) concomitant chronic ischemic and hemorrhagic brain changes, and (4) patency of intracranial vessels. Contrast-enhanced or arterial spin labeling perfusion MRI will be used to (5) measure cerebral perfusion status. Findings from perfusion MRI will be correlated with blood flow information from TCD. MRI including MRA and perfusion sequences will be interpreted centrally in Graz as successfully demonstrated in previous large multicenter stroke studies.
Diagnostic Test: Blood biomarkers — Apart from the assessment of outcome-relevant routine blood parameters of inflammation, coagulation, glucose metabolism, renal and liver function, the investigators will also investigate novel biomarkers of interest that could be indicative of endothelial damage / blood brain barrier disruption. Candidate markers for this purpose are interleukins (i.e., interleukin-6) and matrix metalloproteinases (i.e., MMP-9). Furthermore, the investigators will also measure neurofilament light chain protein as a marker for neuro-axonal damage that has been shown to indicate cerebral tissue destruction including vascular brain lesions with a very high sensitivity.
  For analysis, peripheral blood will be taken by venipuncture on day one and at follow- up three months after MT. Serum will be immediately stored at -80°C according to international consensus guidelines. Markers will be centrally analyzed in the neurological laboratory of the Department of Neurology, Medical University of Graz.

SUMMARY:
Endovascular stroke treatment with mechanical thrombectomy (MT) has become the standard therapy for intracranial large vessel occlusion (LVO). The most serious MT-related complication is secondary intracranial hemorrhage (ICH) occurring in 20-25%. Post- recanalization hyperperfusion might be an important risk factor/mechanism of MT-related ICH. In pilot studies, bedside transcranial Duplex sonography (TCD) was identified as a promising screening tool for cerebral hyperperfusion predicting ICH - the hallmark feature of reperfusion injury.

There is an unmet need to identify risk factors for ICH after MT as it relates to poor prognosis, no proven treatment is available, and it delays/prohibits usage of anticoagulants/-thrombotics necessary for preventing recurrent stroke.

Main objectives:

To explore the range and clinical impact of hemodynamic changes after MT as detected on bedside TCD.

To assess whether patients with increased blood flow velocity in the recanalized middle cerebral artery (MCA) are at a higher risk to develop ICH / vasogenic brain edema (reperfusion injury) after MT.

To investigate if the underlying mechanism is cerebral hyperperfusion (confirmed by perfusion MRI).

To additionally study the role of blood biomarkers of blood-brain-barrier / endothelial dysfunction and neuroaxonal damage on reperfusion injury and short-term prognosis.

Approach / methods:

Prospective, longitudinal Austrian multicentre study conducted at three high-volume stroke centers (Graz, Innsbruck, Salzburg). The investigators will recruit consecutive stroke patients with anterior circulation L VO treated by MT. Immediately after MT, experienced sonographers will perform bedside TCD to determine MCA blood flow status, which will be repeated after 24-48h and on day 7. On day one after MT, brain MRI with perfusion serves to assess infarct size, secondary ICH, (vasogenic) brain edema and perfusion status. MRI will be centrally analyzed in the neuroimaging lab of Graz, blinded to clinical, laboratory and sonographic information. Blood samples for the analysis of biomarkers of endothelial (blood-brain barrier) dysfunction and neuroaxonal damage (neurofilament light) will be taken on day one and at three months post-MT. Neurological outcome will be rated according to the modified Rankin Scale at three months post-stroke.

DETAILED DESCRIPTION:
Endovascular stroke treatment with mechanical thrombectomy (MT) has become the standard therapy for intracranial large vessel occlusion (LVO). The most serious MT-related complication is secondary intracranial hemorrhage (ICH) occurring in 20-25%. Post- recanalization hyperperfusion might be an important risk factor/mechanism of MT-related ICH. In pilot studies, bedside transcranial Duplex sonography (TCD) was identified as a promising screening tool for cerebral hyperperfusion predicting ICH - the hallmark feature of reperfusion injury.

There is an unmet need to identify risk factors for ICH after MT as it relates to poor prognosis, no proven treatment is available, and it delays/prohibits usage of anticoagulants/-thrombotics necessary for preventing recurrent stroke.

Main objectives:

To explore the range and clinical impact of hemodynamic changes after MT as detected on bedside TCD.

To assess whether patients with increased blood flow velocity in the recanalized middle cerebral artery (MCA) are at a higher risk to develop ICH / vasogenic brain edema (reperfusion injury) after MT.

To investigate if the underlying mechanism is cerebral hyperperfusion (confirmed by perfusion MRI).

To additionally study the role of blood biomarkers of blood-brain-barrier / endothelial dysfunction and neuroaxonal damage on reperfusion injury and short-term prognosis.

Approach / methods:

Prospective, longitudinal Austrian multicentre study conducted at three high-volume stroke centers (Graz, Innsbruck, Salzburg). The investigators will recruit consecutive stroke patients with anterior circulation L VO treated by MT. Immediately after MT, experienced sonographers will perform bedside TCD to determine MCA blood flow status, which will be repeated after 24-48h and on day 7. On day one after MT, brain MRI with perfusion serves to assess infarct size, secondary ICH, (vasogenic) brain edema and perfusion status. MRI will be centrally analyzed in the neuroimaging lab of Graz, blinded to clinical, laboratory and sonographic information. Blood samples for the analysis of biomarkers of endothelial (blood-brain barrier) dysfunction and neuroaxonal damage (neurofilament light) will be taken on day one and at three months post-MT. Neurological outcome will be rated according to the modified Rankin Scale at three months post-stroke.

Level of originality:

Human studies on reperfusion injury after MT are lacking. If the investigator's hypothesis would hold true and the investigators could show that cerebral hemodynamic changes after MT would increase the risk for post-interventional intracranial bleeding complications and poor outcome, the investigators would provide an easy-available, repeatable bedside screening and monitoring tool (TCD), which has the potential to guide individualized patient treatment in the early postinterventional period after MT.

The study was registered on Clinicaltrials.gov after start of recruitment.

ELIGIBILITY:
Inclusion Criteria:

* stroke due to large vessel occlusion of the anterior cerebral circulation (internal carotid artery, middle cerebral artery) receiving mechanical thrombectomy.

Exclusion Criteria:

* basilar artery occlusion
* age below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke due to large vessel occlusion of the anterior cerebral circulation (internal carotid artery, middle cerebral artery) receiving mechanical thrombectomy.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Rate of intracranial hemorrhage | Day one after mechanical thrombectomy
  Rate of intracranial hemorrhage (indicator of reperfusion injury) on neuroimaging at day one after mechanical thrombectomy.
Rate of (vasogenic) brain edema | Day one after mechanical thrombectomy
  Rate of (vasogenic) brain edema (indicator of reperfusion injury) on neuroimaging at day one after mechanical thrombectomy.

SECONDARY OUTCOMES:
Cerebral blood flow changes on TCD | Immediately, 24-48 hours and 7 days post-thrombectomy, and after 3 months poststroke
  The range of cerebral blood flow changes on TCD and its correlation with perfusion MRI.
Change of symptomatic intracranial hemorrhage | Immediately, 24-48 hours and 7 days post-thrombectomy.
  Rate of symptomatic intracranial hemorrhage post-thrombectomy.
Inhospital mortality | Median inhospital stay of 7 days
  Early inhospital mortality
Change of functional neurological outcome | Hospital discharge (median of 7 days) and after 3 months poststroke
  Functional neurological outcome (according to the modified Rankin Scale with score of 0-6; higher scores indicating more severe disability) including mortality at three months post-stroke.

CONTACTS AND LOCATIONS:
Locations (3):
- Austria (3):
  - Medical Univerity of Graz, Department of Neurology, Graz, Styria
  - Medical University of Innsbruck, Department of Neurology, Innsbruck, Tyrol
  - Paracelsus Medical University, Department of Neurology, Salzburg